CLINICAL TRIAL: NCT03549572
Title: Validation and Feasibility of the Coma Recovery Scale-Revised for Accelerated Standardized Assessment (CRSR-FAST): a Brief, Standardized Assessment Instrument to Monitor Recovery of Consciousness in the Intensive Care Unit
Brief Title: Validity and Feasibility of the CRSR-FAST
Acronym: CRSR-FAST
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yelena G Bodien, Research Scientist, Massachusetts General Hospital
Other Study IDs: 2015P000147
Record Dates: First submitted 2018-05-25; First posted 2018-06-08 (Actual); Results first posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-08

CONDITIONS: Disorder of Consciousness; Traumatic Brain Injury
MeSH Terms: conditions — Consciousness Disorders; Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Severe Traumatic Brain Injury: We will administer Coma Recovery Scale-Revised (CRS-R) and the Coma Recovery Scale Revised For Accelerated Standardized Testing (CRSR-FAST) to patients in the intensive care unit who have impaired level of consciousness resulting from a severe traumatic brain injury.
  Interventions: Behavioral: Coma Recovery Scale-Revised

INTERVENTIONS:
Behavioral: Coma Recovery Scale-Revised — Patients will be assessed using the CRS-R and the CRSR-FAST. The CRS-R is a standardized neurobehavioral rating scale that consists of 23 items organized into six subscales that address arousal, auditory, visual, motor, oromotor/verbal, and communication systems. Each subscale is organized hierarchically, with lower items representing reflexive behaviors and higher items indicative of cognitively-mediated behaviors. Reliability and validity have been demonstrated in multiple studies. The CRSR-FAST consists of 10 items organized into 4 subscales that address arousal, visual, motor and verbal/oromotor systems. Each subscale is organized hierarchically, with lower items representing reflexive behaviors and higher items indicative of cognitively-mediated behaviors.

SUMMARY:
The CRS-R is a standardized and validated bedside assessment of conscious awareness. It is used routinely for diagnosis and prognosis of patients with disorders of consciousness (DOC) as well as in research settings. One limitation of the CRS-R is the lengthy administration time required to obtain a total score. Administration time can vary from approximately 15-30 minutes, depending on the patient's level of responsiveness. For this reason, the CRS-R is rarely administered in the acute hospital setting. Less time-consuming scales and metrics are used to assess conscious awareness in the acute hospital/ICU setting, but they lack specificity and sensitivity and have not been validated, increasing the potential for misdiagnosis. We have developed the CRSR-FAST and aim to test its validity, inter- and intra- rater reliability. We anticipate that, compared with the CRS-R, the CRSR-FAST will be less time-consuming to administer and score, but will maintain a high level of sensitivity to detecting signs of consciousness in severely brain injured patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Fluent in English
* Surrogate available to provide informed consent
* History of severe acquired brain injury
* Sustained a traumatic brain injury (TBI, defined by damage to brain tissue caused by an external mechanical force),
* Be within 3 weeks of injury
* Have a total Glasgow Outcome Scale (GCS) score <9 within the first 48 hours of injury,
* Be unable to follow simple commands consistently at the time of enrollment

Exclusion Criteria:

* History of developmental, neurologic, or major psychiatric disorder resulting in ongoing functional disability up to the time of the current injury
* Physician orders for comfort measures only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll adults with a impaired level of consciousness resulting from severe traumatic brain injury who are recovering in the intensive care unit.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-08-28 (Actual); Primary Completion 2022-12-04 (Actual); Study Completion 2022-12-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giacino JT, Kalmar K, Whyte J. The JFK Coma Recovery Scale-Revised: measurement characteristics and diagnostic utility. Arch Phys Med Rehabil. 2004 Dec;85(12):2020-9. doi: 10.1016/j.apmr.2004.02.033. PMID 15605342

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Severe Traumatic Brain Injury
Started | 56
Completed | 45
Not Completed | 11

BASELINE CHARACTERISTICS:
Groups:
- Severe Traumatic Brain Injury: We will administer Coma Recovery Scale-Revised (CRS-R) and the Coma Recovery Scale Revised For Accelerated Standardized Testing (CRSR-FAST) to patients in the intensive care unit who have impaired level of consciousness resulting from a severe traumatic brain injury.
  Coma Recovery Scale-Revised: Patients will be assessed using the CRS-R and the CRSR-FAST. The CRS-R is a standardized neurobehavioral rating scale that consists of 23 items organized into six subscales that address arousal, auditory, visual, motor, oromotor/verbal, and communication systems. Each subscale is organized hierarchically, with lower items representing reflexive behaviors and higher items indicative of cognitively-mediated behaviors. Reliability and validity have been demonstrated in multiple studies. The CRSR-FAST consists of 5 items that address visual, motor and verbal/oromotor systems.
Arm/Group | Severe Traumatic Brain Injury
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 35
  >=65 years | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 40
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 45

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Agreement
Description: Diagnostic agreement between the Coma Recovery Scale-Revised (CRS-R) and the CRSR For Accelerated Standardized Testing (CRSR-FAST). The CRS-R is a standardized neurobehavioral rating scale used to monitor recovery of consciousness. Total scores on the CRS-R range from 0 to 23 with high scores generally indicating greater recovery. Six subscales on the CRS-R are summed to provide the total score: auditory function, visual function, motor function, oromotor/verbal function, communication and arousal. Evidence of specific behaviors on these subscales provides a diagnosis of vegetative state, minimally conscious state (MCS), or emerged from MCS. The CRSR-FAST is an abbreviated version of the CRS-R. We tested concurrent validity by comparing CRS-R and CRSR-FAST diagnostic ratings using the simple kappa coefficient; values close to 0 indicate no agreement and values close to 1 indicate almost perfect agreement. We established an a priori threshold of ≥ 0.60 to indicate substantial validity
Time Frame: 48 hours
Measure: Number; unit: Simple Kappa (SE)
Arm/Group | Severe Traumatic Brain Injury
Number analyzed (Participants) | 45
Simple Kappa (SE) | .68

2. Other Pre Specified Outcome: CRSR-FAST Test-Retest Reliability
Description: CRSR-FAST test-retest reliability using Mak's ρ. The CRSR-FAST was administered twice by 2 blinded raters. Mak's ρ values close to 0 indicate no agreement and values close to 1 indicate almost perfect reliability. We established an a priori threshold of ≥ 0.60 to indicate substantial reliability
Time Frame: 48 hours
Measure: Number; unit: Mak's ρ
Arm/Group | Severe Traumatic Brain Injury
Number analyzed (Participants) | 45
Mak's ρ | 0.76

3. Other Pre Specified Outcome: CRSR-FAST Interrater Reliability
Description: CRSR-FAST interrupter reliability using Mak's ρ. The CRSR-FAST was administered twice by the same rater. Mak's ρ values close to 0 indicate no agreement and values close to 1 indicate almost perfect reliability. We established an a priori threshold of ≥ 0.60 to indicate substantial reliability
Time Frame: 48 hours
Measure: Number; unit: Mak's ρ
Arm/Group | Severe Traumatic Brain Injury
Number analyzed (Participants) | 45
Mak's ρ | 0.91

ADVERSE EVENTS:
Time Frame: 48 hours
Description: This is an observational study with no intervention.
Groups:
- Severe Traumatic Brain Injury: We will administer Coma Recovery Scale-Revised (CRS-R) and the Coma Recovery Scale Revised For Accelerated Standardized Testing (CRSR-FAST) to patients in the intensive care unit who have impaired level of consciousness resulting from a severe traumatic brain injury.
  Coma Recovery Scale-Revised: Patients will be assessed using the CRS-R and the CRSR-FAST. The CRS-R is a standardized neurobehavioral rating scale that consists of 23 items organized into six subscales that address arousal, auditory, visual, motor, oromotor/verbal, and communication systems. Each subscale is organized hierarchically, with lower items representing reflexive behaviors and higher items indicative of cognitively-mediated behaviors. Reliability and validity have been demonstrated in multiple studies. The CRSR-FAST consists of 10 items organized into 4 subscales that address arousal, visual, motor and verbal/oromotor systems. Each subscale is organized hierarchically, with lower items representing reflexive behaviors and higher items indicative of cognitively-mediated behaviors.
  There were no adverse events.
Arm/Group | Severe Traumatic Brain Injury
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

LIMITATIONS AND CAVEATS:
The full-length CRS-R was administered only one time while the CRSR-FAST was administered 3 times. Fluctuations in level of consciousness over 48 hours may have affected the full-length CRS-R assessment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-08): https://cdn.clinicaltrials.gov/large-docs/72/NCT03549572/Prot_SAP_000.pdf